CLINICAL TRIAL: NCT01853995
Title: Class II Division 1 Malocclusions Treated With Fixed Lingual Mandibular Growth Modificator (FLMGM): The Mechanism of Sagittal Occlusal Correction
Brief Title: Mechanism of Class II Correction With Fixed Lingual Mandibular Growth Modificator (FLMGM)
Acronym: FLMGM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Principal Investigator, Osama AlAli, Dr., Damascus University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLMGM: Mechanism of Correction
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Class II Division 1 Malocclusion
Keywords: Fixed Lingual Mandibular Growth Modificator (FLMGM); Class II division 1 malocclusion; Sagittal Occlusal Correction; Skeletal changes; Dental changes
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FLMGM Treatment Group (Experimental): Cl II/1 patients treated with Fixed Lingual Mandibular Growth Modificator (FLMGM)
  Interventions: Device: Fixed Lingual Mandibular Growth Modificator (FLMGM)
- Untreated Class II Control Group (No Intervention): control group

INTERVENTIONS:
Device: Fixed Lingual Mandibular Growth Modificator (FLMGM) — New Class II Corrector
  Other Names: Fixed Lingual Mandibular Growth Modification Appliance
  Arms: FLMGM Treatment Group

SUMMARY:
The aim of the current controlled trial was to assess the possible net skeletal and dental effects of FLMGM treatment in relation to growth with emphasis on the contribution of skeletal and dental changes to sagittal correction of Cl II/1 malocclusion.

The null hypothesis stated that there were no significant differences in dentoskeletal changes between FLMGM treated group and control untreated group.

DETAILED DESCRIPTION:
The current study was prospective, controlled, parallel groups, clinical trial conducted at the department of Orthodontics between May 2009 and June 2011. The protocol of study was approved by the council of scientific research and postgraduate studies, on the 5/April/2009.

Of the 43 patients initially enrolled, 38 completed this trial and comprised the final sample, and 5 (4 treated, 1 untreated) were excluded.

The final sample comprised 38 subjects who completed this trial. All patients and parents gave prior informed consent to their inclusion in the investigation.

Patients of both groups were followed on a parallel basis during a period of 8 months and the trial included all patients regardless of achievement of a Class I incisor relationship. All patient of treatment group (n=21) were treated using FLMGM without extractions or any other form of orthodontic treatment, though the treatment was continued beyond this time point if the Class II malocclusion was not fully corrected and clinical objectives were not achieved. On the other hand, no orthodontic treatment was performed during that duration for the subjects of control group (n=17), and most of control subjects were offered suitable treatment at a later date.

For each patient, a direct digital lateral cephalogram was taken pre- and post- treatment/observation using PAX 400 (VATECH CO., Korea) with the same settings. All cephalograms were digitized on screen by a cursor-driven mouse and analyzed in a blind manner by the same orthodontist using a commercial cephalometric software (Viewbox, version 3.1.1.13, dHAL Software, Kifissia , Hellas, Greece). All measurements were reduced to life size (radiographic enlargement of 7.54 % in the median plane).

At the end of the treatment/observation period, sagittal occlusal (SO) analysis, according to the method of Pancherz modified by Franchi et al, was applied to assess sagittal occlusal changes and identify the mechanism of Class II correction. Moreover, the total mandibular length (Condyle-Gnathion) was measured.

The sample was used as a whole and not differentiated by sex. Pretreatment equivalence and comparison of changes observed in the FLMGM and control groups were tested for significance with independent-sample t-test using SPSS, version 16.0. Changes occurring during the examination period in each group were tested with paired-sample t-test. P values of less than 0.05 were considered statistically significant.

To assess the method error, twenty cephalograms were picked at random from the treatment and control groups and redigitized and analyzed by the same orthodontist after an interval of 1 month, and the combined error of cephalometric method was calculated by Dahlberg's formula.

ELIGIBILITY:
Inclusion Criteria:

* Cl II/1 malocclusion with an overjet greater than 4 mm.
* Mild to moderate Class II Skeletal pattern (A-N-B > 4°) with retrognathic mandible (S-N-B < 76°).
* Growth potential. Fishman skeletal maturation indicator (SMI) method was used to assess the hand-wrist radiographs, and only patients in the peak of the pubertal growth spurt, which occurs on average between SMIs 4 to 7, at the beginning of the treatment/observation period were invited.

Exclusion Criteria:

* craniofacial syndromes
* clinically obvious facial asymmetry
* extreme vertical disproportion
* prior orthodontic therapy
* permanent tooth extractions
* significant medical history

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Overjet reduction and Class II molar correction | 8 months

SECONDARY OUTCOMES:
Total mandibular length (Co-Gn) | 8 months

OTHER OUTCOMES:
Standard Dental and skeletal changes | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Osama H Alali, PhD, Principal Investigator — Senior Lecturer, Department of Orthodontics, School of Dentistry, University of Aleppo, Syria
Locations (1):
- Department of Orthodontics, School of Dentistry, University of Damascus, Damascus, Rif-dimashq Governorate, Syria